CLINICAL TRIAL: NCT06970223
Title: Phase 1, Open-Label, Randomised Crossover Study Assessing the Tolerability and Acceptability of Long Acting Cabotegravir Intramuscular and Lenacapavir Subcutaneous Injections Over Time in Healthy Adults Without HIV
Brief Title: A Study to Investigate if Long Acting Cabotegravir (CAB) and Lenacapavir (LEN) Injections Are Tolerable and Acceptable When Administered to Healthy Adults Without HIV
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 223616
Record Dates: First submitted 2025-04-11; First posted 2025-05-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
Keywords: Long-acting; Tolerability; Acceptability; Injection site reactions; Cabotegravir; Lenacapavir; Healthy adults
MeSH Terms: conditions — HIV Infections; Injection Site Reaction | interventions — cabotegravir

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAB LA/LEN LA Group (Experimental): Participants receive the CAB LA injection at Day 1 followed by the LEN LA injections at Day 15.
  Interventions: Drug: Cabotegravir long-acting; Drug: Lenacapavir long-acting
- LEN LA/CAB LA Group (Experimental): Participants receive the LEN LA injections at Day 1 followed by the CAB LA injection at Day 15.
  Interventions: Drug: Cabotegravir long-acting; Drug: Lenacapavir long-acting

INTERVENTIONS:
Drug: Cabotegravir long-acting — A single CAB LA injection administered intramuscularly.
  Other Names: Cabotegravir
Drug: Lenacapavir long-acting — Two LEN LA injections administered subcutaneously.

SUMMARY:
This study will evaluate the tolerability and acceptability of injection site reactions (ISRs) of two long-acting (LA) injectables. Additional characteristics of the ISRs will be investigated and described as well as safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply:

1. At the time of obtaining informed consent, 18 years of age.
2. Body weight 50 kg and BMI within the range 18 to 32 kg/m2 (inclusive).
3. Participants who are overtly healthy as determined by medical evaluation by a responsible and experienced physician, including medical history, physical examination, laboratory tests and cardiac monitoring.
4. A participant with a significant clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included if the investigator determines and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. A single repeat of a procedure or lab parameter is allowed to determine eligibility.
5. Male or female at birth (transgender individuals are not excluded but LEN may interfere with gender affirming hormones including increasing thrombotic risk. This should be discussed with Medical Monitor).
6. All participants are expected to use barrier methods for HIV/STI prevention and should be counselled accordingly at all visits.
7. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
8. Participants assigned female at birth are eligible to participate if they are not pregnant or breast/chest-feeding, and at least 1 of the following conditions applies:

   * Is not a person of childbearing potential (POCBP) OR
   * Is a POCBP and using a contraceptive method that is highly effective, with a failure rate of <1%. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.
9. A POCBP must have a negative highly sensitive pregnancy test (urine and/or serum as required) within the 21 days before the dose of study intervention.
10. Must be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data. The investigator may contact the ViiV healthcare (VH) medical monitor to discuss the inclusion of participants who have a history of specific conditions that are not expected to interfere with their participation in the study.
2. Suspected or known active, serious infection(s).
3. Abnormal blood pressure as determined by the investigator.
4. History of any malignancy within the past 5 years. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy which is considered cured with minimal risk of recurrence. Participants under evaluation for possible malignancy are not eligible.
5. Breast cancer within the past 10 years
6. Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
7. The participant has an underlying skin disease or disorder (i.e., infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) that would interfere with assessment of injection sites.
8. Current or anticipated need for chronic anti-coagulation.
9. Participants considered to have insufficient musculature to allow safe intramuscular (e.g., gluteus medius, vastus lateralis) or sufficient subcutaneous thickness to allow subcutaneous administration in the opinion of the investigator.
10. Any Positive Treponeme Specific Serologic testing (positive T. Pallidum antibody immunoassay + Rapid plasma reagin [RPR] or positive T. Pallidum antibody immunoassay + Treponema pallidum particle agglutination [TPPA]) is exclusionary.
11. Presence of HBsAg, or positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of study treatment.
12. Have a history of osteoporosis or bone fragility fractures.
13. Participants who, in the investigator's judgment, poses a significant suicidality risk. Participant's history of suicidal behaviour and/or suicidal ideation should be considered when evaluating for suicide risk.
14. Any preexisting physical or mental condition which, in the opinion of the Investigator or the Medical Monitor, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
15. Participants receiving any protocol-prohibited medication and who are unwilling or unable to switch to an alternate medication.
16. Treatment with any of the following agents within 60 days of screening: radiation therapy, cytotoxic chemotherapeutic agents, any systemic immune suppressant.
17. Past or intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing.
18. Use of glucocorticoids (through any route).
19. Exposure to more than 4 new investigational products within 12 months prior to the first dosing day.
20. Current enrolment or past participation in another investigational study in which an investigational intervention (e.g., drug, human blood product, monoclonal antibody, vaccine, invasive device) was administered within 1 month, 5 half-lives or twice the duration of the biological effect of the test agent prior to screening (whichever is longer).
21. Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in the study of an investigational compound.
22. Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 triglycerides or lipid abnormalities. A single repeat test is allowed during the screening period to verify a result.
23. ALT greater than or equal to (>=) 1.5x ULN. A single repeat test is allowed within a single Screening period to determine eligibility.
24. Total bilirubin >=1.5x ULN (isolated total bilirubin greater than [>] 1.5xULN is acceptable if total bilirubin is fractionated and direct bilirubin less than [<] 35%). A single repeat test is allowed within a single screening period to determine eligibility.
25. Creatinine clearance (eGFR) of <60 mL/min/1.73 m2 via CKD-EPI method.
26. Positive HIV antibody/antigen test (HIV-1, HIV-2) at screening or enrolment. Participants will be advised regarding safer sex. In the event a participant acquires HIV during the study they will be required to withdraw from the study and will be referred urgently to an HIV treatment center for further management.
27. Clinically significant cardiovascular disease, as defined by history/evidence of congestive heart failure, symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting surgery or percutaneous transluminal coronary angioplasty or any clinically significant cardiac disease.
28. Grade 3 or Grade 4 proteinuria or glycosuria at screening that is unexplained or not clinically manageable.
29. Participant is unlikely to adhere to the study procedures, keep appointments, is planning to relocate during the study, or remain on study through to its conclusion.
30. Alcohol or substance use that, in the opinion of the study investigator and medical monitor, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records).
31. Participant has an implant/enhancement (including fillers) at the area of proposed injection; or tattoo or other dermatological condition overlying the area for IM or SC injection (e.g., gluteus medius, vastus lateralis or anterior abdominal wall) or any other area which may significantly interfere with interpretation of injection site reactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting very acceptable or totally acceptable local reactions | 7 days after each injection (injections administered on Day 1 and Day 15)
  The analysis is performed using the 21-item perception of injection (PIN) questionnaire which includes 21 items grouped into 4 multi-item domains: 'Acceptance of ISR' scale score (2 items); 'Bother from ISR' scale score (6 items); 'Leg movement' scale score (4 items); 'Sleep' scale score (4 items); and 5 standalone items: pain during injection; anxiety before injection; anxiety after injection; willingness to be injected in the future; and overall satisfaction with mode of administration. Participant responses are scored on a 5-point Likert scale, where 1 represents the least favorable perception of injection and 5 the most favorable, with domain scores calculated as the mean of all items in that domain.
  "Acceptance of ISR" is reported in this outcome measure for 2 scores: "very acceptable ISR: and "totally acceptable ISR".

SECONDARY OUTCOMES:
Percentage of participants reporting very acceptable or totally acceptable local reactions at days 43 and 190 | At Day 43 (28 days after second injection) and Day 190 (26 weeks after second injection)
  The analysis is performed using the 21-item PIN questionnaire which includes 21 items grouped into 4 multi-item domains: 'Acceptance of ISR' scale score (2 items); 'Bother from ISR' scale score (6 items); 'Leg movement' scale score (4 items); 'Sleep' scale score (4 items); and 5 standalone items: pain during injection; anxiety before injection; anxiety after injection; willingness to be injected in the future; and overall satisfaction with mode of administration. Participant responses are scored on a 5-point Likert scale, where 1 represents the least favorable perception of injection and 5 the most favorable, with domain scores calculated as the mean of all items in that domain.
  "Acceptance of ISR" is reported in this outcome measure for 2 scores: "very acceptable ISR: and "totally acceptable ISR".
Mean injection site reaction scores, over time, post-injection, at days 8 and 22 | At Day 8 and Day 22 (7 days after each injection visit)
  The analysis is performed using the 21-item PIN questionnaire which includes 21 items grouped into 4 multi-item domains: 'Acceptance of ISR' scale score (2 items); 'Bother from ISR' scale score (6 items); 'Leg movement' scale score (4 items); 'Sleep' scale score (4 items); and 5 standalone items: pain during injection; anxiety before injection; anxiety after injection; willingness to be injected in the future; and overall satisfaction with mode of administration. Participant responses are scored on a 5-point Likert scale, where 1 represents the least favorable perception of injection and 5 the most favorable, with domain scores calculated as the mean of all items in that domain.
Median injection site reaction scores, over time, post-injection, at days 8 and 22 | At Day 8 and Day 22 (7 days after each injection visit)
  The analysis is performed using the 21-item PIN questionnaire which includes 21 items grouped into 4 multi-item domains: 'Acceptance of ISR' scale score (2 items); 'Bother from ISR' scale score (6 items); 'Leg movement' scale score (4 items); 'Sleep' scale score (4 items); and 5 standalone items: pain during injection; anxiety before injection; anxiety after injection; willingness to be injected in the future; and overall satisfaction with mode of administration. Participant responses are scored on a 5-point Likert scale, where 1 represents the least favorable perception of injection and 5 the most favorable, with domain scores calculated as the mean of all items in that domain.
Mean injection site reaction scores, over time, post-injection, at days 43 and 190 | At Day 43 (28 days after second injection) and Day 190 (26 weeks after second injection)
  The analysis is performed using the 21-item PIN questionnaire which includes 21 items grouped into 4 multi-item domains: 'Acceptance of ISR' scale score (2 items); 'Bother from ISR' scale score (6 items); 'Leg movement' scale score (4 items); 'Sleep' scale score (4 items); and 5 standalone items: pain during injection; anxiety before injection; anxiety after injection; willingness to be injected in the future; and overall satisfaction with mode of administration. Participant responses are scored on a 5-point Likert scale, where 1 represents the least favorable perception of injection and 5 the most favorable, with domain scores calculated as the mean of all items in that domain.
Median injection site reaction scores, over time, post-injection, at days 43 and 190 | At Day 43 (28 days after second injection) and Day 190 (26 weeks after second injection)
  The analysis is performed using the 21-item PIN questionnaire which includes 21 items grouped into 4 multi-item domains: 'Acceptance of ISR' scale score (2 items); 'Bother from ISR' scale score (6 items); 'Leg movement' scale score (4 items); 'Sleep' scale score (4 items); and 5 standalone items: pain during injection; anxiety before injection; anxiety after injection; willingness to be injected in the future; and overall satisfaction with mode of administration. Participant responses are scored on a 5-point Likert scale, where 1 represents the least favorable perception of injection and 5 the most favorable, with domain scores calculated as the mean of all items in that domain.
Change in the intensity of post-injection site pain assessed over time | At days 1, 2, 5 and 8 for the first injection and days 15, 16, 19, and 22 for the second injection
  The analysis is performed using the numerical rating scale (NRS), which is a visual analogue scale that assesses the maximum level of pain experienced with injections ranging from 0 (no pain) to 10 (extreme pain). An NRS related to each injection is self-administered electronically at the clinic visits at the same timepoints after each injection
Percentage of participants with ISRs overall and by severity | Up to 6 months post any injection
  The ISRs severity is graded using the Division of Acquired Immunodeficiency Syndrome (DAIDS) criteria Version 2.1 where grades are defined based on numeric criteria as follows Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: potentially life-threatening. A higher grade indicates greater severity.
Percentage of participants with specific ISRs of interest | Up to 6 months post any injection
  The ISRs of interest are nodules (maximum diameter and visibility over time), pigmentation changes (assessed surface area, distinction of hyperpigmentation vs hypopigmentation), and induration/ swelling (visibility over time).
Mean duration of ISRs | Up to 6 months post any injection
Median duration of ISRs | Up to 6 months post any injection
Percentage of participants with adverse events (AEs) overall and by severity | Up to 6 months post a single dose of CAB LA and LEN LA sequentially administered
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. The AEs severity is graded using the DAIDS criteria Version 2.1 where grades were defined based on numeric criteria as follows Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: potentially life-threatening. A higher grade indicates greater severity.
Number of participants with laboratory abnormalities | Up to 6 months post any injection
Number of participants with change in laboratory parameters over time | Up to 6 months post any injection compared to Baseline (Day 1)
Maximum change in toxicity grade from baseline in laboratory values | Up to 6 months post any injection compared to Baseline (Day 1)
  Toxicity is graded using the DAIDS criteria Version 2.1 where grades were defined based on numeric criteria as follows Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: potentially life-threatening. A higher grade indicates greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.ViiV-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.ViiV-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf